CLINICAL TRIAL: NCT01680770
Title: Use of Ultrasonography to Determine Fluid-responsiveness for Shock in a Population of Intensive Care Unit Patients
Status: Active, not recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 10-566B
Record Dates: First submitted 2012-06-18; First posted 2012-09-07 (Estimated); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Hypotension
Keywords: shock; transthoracic echocardiography; critical care
MeSH Terms: conditions — Hypotension; Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Hypotensive patients in shock

SUMMARY:
The objective of our study is to determine the correlation of transthoracic ultrasonographic indices of fluid responsiveness to changes in direct measures of cardiac output and to compare them to other established predictors of fluid responsiveness such as central venous pressure variation, systolic arterial pressure variation and pulse pressure variation in a broad population of patients.

Hypothesis: There will be a significant difference in the inferior vena cava respiratory variation and subclavian vein respiratory variation between responders and non-responders to intravenous fluid challenge in a broad population of patients with shock.

DETAILED DESCRIPTION:
Shock is a common occurrence in the intensive care unit (ICU), and the management of this condition frequently requires the administration of intravenous fluids (IVF). Multiple studies have shown that only about 50% of these patients will respond to fluids. The ability to predict which patients will respond is an important tool for clinicians to treat shock while avoiding unnecessary fluid administration in those who are unlikely to respond. This is essential to avoid the adverse effects of fluid loading that can occur.

A number of studies have attempted to determine predictors of volume-responsiveness through various methods, including the use of ultrasonography performed by intensivists, anesthesiologists and emergency medicine physicians. The currently published studies establish predictors of fluid-responsiveness in their populations. However, there has been large variability in the study designs, making it difficult to compare different modalities.

The objective of our study is to determine the correlation of transthoracic ultrasonographic indices of fluid responsiveness to changes in direct measures of cardiac output and to compare them to other established predictors of fluid responsiveness such as central venous pressure variation, systolic arterial pressure variation and pulse pressure variation. Furthermore, we wish to include a broad range of patients with different types of shock in order to determine the generalized applicability of these indices. Additionally, reported success of intensivist-obtained echocardiographic images varies widely in the literature, but most studies do not report which views are most accessible. We plan to study prospectively which views are obtainable and correlate them to patient characteristics.

This would potentially establish echocardiography by an intensivist as a widely applicable, non-invasive, and easily accessible method for determining fluid-responsiveness in a patient with shock. Achievement of this goal would allow clinicians to quickly identify those patients that would respond to fluids and at the same time minimize the administration of fluids to those in whom it is unlikely to benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (> 18 years old) admitted to the intensive care unit.
2. Decision by clinicians to give intravenous fluids for volume expansion.
3. Decision by clinicians to obtain central venous access.

Exclusion Criteria:

1. Patients with known chronic right heart failure syndromes.
2. Patients with terminal conditions in whom aggressive care will not be pursued.
3. Patients with a history of left bundle branch block.
4. Patients will not be excluded on the basis of sex, race, or ethnicity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Intensive Care Unit Patients
Sampling Method: Non-Probability Sample
Enrollment: 124 (Estimated)
Dates: Start 2010-06; Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Fluid Responder vs. Non-responder | pre-fluid challenge baseline and post-fluid challenge (approximately 1 hour)
  Patients will be divided into responder and non-responder groups based on an increase in cardiac output of greater than or equal to 15% as measured by thermodilution from a right heart catheter in response to a one liter normal saline fluid bolus.

SECONDARY OUTCOMES:
Inferior vena cava diameter and respiratory variation | pre-fluid challenge baseline and post-fluid challenge (approximately 1 hour)
  pre-fluid Inferior vena cava diameter and Inferior vena cava respiratory variations will be correlated to fluid responsiveness
subclavian vein diameter and respiratory variation | pre-fluid challenge baseline and post-fluid challenge (approximately 1 hour)
  pre-fluid subclavian diameter and subclavian respiratory variations will be correlated to fluid responsiveness
pulse pressure variation | pre-fluid challenge baseline and post-fluid challenge (approximately 1 hour)
  pre-fluid pulse pressure variation will be correlated to fluid responsiveness
central venous pressure (CVP) and CVP respiratory variation | pre-fluid challenge baseline and post-fluid challenge (approximately 1 hour)
  pre-fluid CVP and CVP respiratory variations will be correlated to fluid responsiveness
pulmonary capillary wedge pressure (PCWP) and respiratory variations of PCWP | pre-fluid challenge baseline and post-fluid challenge (approximately 1 hour)
  pre-fluid PCWP and PCWP respiratory variations will be correlated to fluid responsiveness
Possible views of echocardiogram | pre-fluid challenge baseline and post-fluid challenge (approximately 1 hour)
  Determine percentage of which echocardiographic views are obtainable in a broad population of patients with shock and correlate to patient characteristics
Concurrence with cardiologist interpretation | pre-fluid challenge baseline and post-fluid challenge (approximately 1 hour)
  Determine the rate at which cardiologist concurs with intensivist interpretation of echocardiographic images.

CONTACTS AND LOCATIONS:
Overall Officials: Kress P John, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No